CLINICAL TRIAL: NCT00042094
Title: A Phase 1 Study of Reactogenicity, Safety, Immunogenicity, and Pock Lesion Formation (Take Rate) of a Cell-Cultured Smallpox Vaccine (CCSV) Compared to a Calf Lymph Vaccine (Dryvax®)
Brief Title: Study of Reactogenicity, Safety, Immunogenicity, and Pock Lesion Formation of a Cell-Cultured Smallpox Vaccine Compared to Dryvax®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DynPort Vaccine Company LLC, A GDIT Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SMPX-001
Record Dates: First submitted 2002-07-23; First posted 2002-07-26 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Smallpox
Keywords: Smallpox; Smallpox Vaccine; Vaccinia
MeSH Terms: conditions — Smallpox; Vaccinia

INTERVENTIONS:
Biological: Cell-Cultured Smallpox Vaccine compared to Dryvax®

SUMMARY:
This study will evaluate the safety and efficacy of both Dryvax® and the new cell-cultured vaccine (CCSV) in a comparative fashion. Across 3 cohorts, 150 vaccinia-naive volunteers will be randomly assigned to receive either CCSV (100 volunteers) or Dryvax® (50 volunteers) in a blinded fashion. Subjects will be followed closely for up to 6 months and a subgroup of volunteers will be followed up to 3 years in order to evaluate the duration of immunity following vaccination. Another cohort will enroll 100 vaccinia-experienced volunteers and randomly assign them to receive either CCSV (50 volunteers) or Dryvax® (50 volunteers) and a sub group will be followed up to 3 years. A fifth cohort will enroll 100 vaccinia-naive volunteers and randomly assign them to receive different dilutions of CCSV (1:1, 1:5, 1:25, and 1:50).

ELIGIBILITY:
* Have never received smallpox vaccine or previously received an experimental smallpox vectored vaccine (for vaccinia-naive cohorts only)
* Have been previously vaccinated within the last 10 years (vaccinia-experienced cohort only)
* Must agree to have blood samples banked for future research testing
* Have not participated in any clinical trial using investigational product within past month
* No current or past history of exfoliative skin problems
* Not have regular contact with children under 3 years of age until scab at site of vaccination has fallen off (around 21 days or 3 weeks after vaccination)
* Do not have a positive test for HIV virus, hepatitis C virus, or hepatitis B surface antigen
* Are not a health care worker caring for newborns, patients that are immunocompromised or have skin that is adversely altered
* Will not engage in direct patient care until immunization scab falls off (around 21 days or 3 weeks after vaccination) if health care worker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2002-03; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States